CLINICAL TRIAL: NCT03600805
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Sarilumab in Patients With Giant Cell Arteritis
Brief Title: Evaluation of Efficacy and Safety of Sarilumab in Patients With GCA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Protracted recruitment timeline exacerbated by COVID-19 pandemic
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15068; 2017-002988-18 (EudraCT Number); U1111-1200-2184 (Other: UTN)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — sarilumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo+52 Week Taper (Experimental): Participants received sarilumab-matching placebo as subcutaneous (SC) injection every 2 weeks (q2w) up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone/prednisone-matching placebo tapering oral daily doses for 52 weeks.
  Interventions: Drug: Sarilumab matching placebo; Drug: Prednisone; Drug: Prednisone matching placebo
- Placebo+26 Week Taper (Experimental): Participants received sarilumab-matching placebo as SC injection q2w up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone-matching placebo from Week 26 up to Week 52.
  Interventions: Drug: Sarilumab matching placebo; Drug: Prednisone; Drug: Prednisone matching placebo
- Sarilumab 150mg q2w+26 Week Taper (Placebo Comparator): Participants received sarilumab 150 milligrams (mg) as SC injection q2w up to 52 weeks along with prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone-matching placebo from Week 26 up to Week 52.
  Interventions: Drug: Sarilumab SAR153191; Drug: Prednisone; Drug: Prednisone matching placebo
- Sarilumab 200mg q2w+26 Week Taper (Placebo Comparator): Participants received sarilumab 200 mg as SC injection q2w up to 52 weeks along with prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone-matching placebo from Week 26 up to Week 52.
  Interventions: Drug: Sarilumab SAR153191; Drug: Prednisone; Drug: Prednisone matching placebo

INTERVENTIONS:
Drug: Sarilumab SAR153191 — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Sarilumab 150mg q2w+26 Week Taper; Sarilumab 200mg q2w+26 Week Taper
Drug: Sarilumab matching placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo+26 Week Taper; Placebo+52 Week Taper
Drug: Prednisone — Pharmaceutical form: tablets or capsules Route of administration: oral administration
Drug: Prednisone matching placebo — Pharmaceutical form: capsules Route of administration: oral administration

SUMMARY:
Primary Objective:

To evaluate the efficacy of sarilumab in participants with giant cell arteritis (GCA) as assessed by the proportion of participants with sustained remission for sarilumab compared to placebo, in combination with a corticosteroid (CS) tapering course.

Secondary Objective:

* To demonstrate the efficacy of sarilumab in participants with GCA compared to placebo, in combination with CS taper with regards to:
* Clinical responses (such as responses based on disease remission rates, time to first disease flare) over time.
* Cumulative CS (including prednisone) exposure.
* To assess the safety (including immunogenicity) and tolerability of sarilumab in participants with GCA.
* To measure sarilumab serum concentrations in participants with GCA.
* To assess the effect of sarilumab on sparing glucocorticoid toxicity as measured by glucocorticoid toxicity index (GTI).

DETAILED DESCRIPTION:
Study duration per participant was approximately 82 weeks, including an up to 6-week screening period, 52-week treatment period, and 24-week follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of GCA according to European League Against Rheumatism/American College of Rheumatology classification criteria.
* New onset active disease or refractory active disease.
* At least one of the symptoms of GCA within 6 weeks of baseline.
* Either erythrocyte sedimentation rate greater than or equal to (>=) 30 millimeter per hour or C-reactive protein >=10 mg per liter within 6 weeks of baseline.
* Received or were able to receive prednisone 20-60 mg/day for the treatment of active GCA.

Exclusion criteria:

* Organ transplantation recipient (except corneas, unless it is within 3 months prior to baseline visit).
* Major ischemic event, unrelated to GCA, within 12 weeks of screening.
* Any prior use of the following therapies, for the treatment of GCA:
* Janus kinase inhibitor (e.g., tofacitinib) within 4 weeks of baseline.
* Cell-depletion agents (e.g., anti CD20) without evidence of recovery of B cells to baseline level.
* Abatacept within 8 weeks of baseline.
* Anakinra within 1 week of baseline.
* Tumor necrosis factor inhibitors within 2-8 weeks (etanercept within 2 weeks; infliximab, certolizumab, golimumab, or adalimumab within 8 weeks), or less than at least 5 half-lives had elapsed prior to baseline, whichever was longer.
* Therapeutic failure, including inadequate response or intolerance, or contraindication, to biological Interleukin 6 (IL-6) IL-6/(R) antagonist (prior experience with IL-6/(R) antagonist that was terminated for reasons unrelated to therapeutic failure at least 3 months before baseline was not exclusionary).
* Use of any alkylating agents including cyclophosphamide within 6 months of baseline.
* Use of immunosuppressant, such as hydroxychloroquine, cyclosporine, azathioprine, mycophenolate mofetil or leflunomide within 4 weeks of baseline. (Use of methotrexate (MTX) not exceeding 25 mg per week and had been stable for at least 3 months prior to baseline was not exclusionary).
* Concurrent use of systemic CS for conditions other than GCA.
* Use of intervascular CS at a dose equivalent to 100 mg of methylprednisolone or higher within 8 weeks of baseline for GCA therapy.
* Pregnant or breastfeeding woman.
* Participants with active or untreated latent tuberculosis.
* Participants with history of invasive opportunistic infections.
* Participants with fever associated with infection or chronic, persistent or recurring infections requiring active treatment.
* Participants with uncontrolled diabetes mellitus.
* Participants with non-healed or healing skin ulcers.
* Participants who received any live, attenuated vaccine within 3 months of baseline.
* Participants who are positive for hepatitis B, hepatitis C and/or HIV.
* Participants with a history of active or recurrent herpes zoster.
* Participants with a history of or prior articular or prosthetic joint infection.
* Prior or current history of malignancy.
* Participants who have had surgery within 4 weeks of screening or planned surgery during study.
* Participants with a history of inflammatory bowel disease or severe diverticulitis or previous gastrointestinal perforation..

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (61):
- United States (6):
  - Investigational Site Number 8400002, Boca Raton, Florida
  - Investigational Site Number 8400017, Gainesville, Florida
  - Investigational Site Number 8400014, Iowa City, Iowa
  - Investigational Site Number 8400018, Portland, Oregon
  - Investigational Site Number 8400019, Philadelphia, Pennsylvania
  - Investigational Site Number 8400011, Dallas, Texas
- Argentina (2):
  - Investigational Site Number 0320001, Buenos Aires
  - Investigational Site Number 0320002, Caba
- Australia (3):
  - Investigational Site Number 0360003, Camberwell
  - Investigational Site Number 0360006, Clayton
  - Investigational Site Number 0360001, Kogarah
- Investigational Site Number 0560001, Leuven, Belgium
- Canada (5):
  - Investigational Site Number 1240007, Hamilton
  - Investigational Site Number 1240010, Montreal
  - Investigational Site Number 1240001, Rimouski
  - Investigational Site Number 1240005, Sherbrooke
  - Investigational Site Number 1240003, Trois-Rivières
- Investigational Site Number 1910001, Zagreb, Croatia
- Denmark (2):
  - Investigational Site Number 2080002, Aarhus C
  - Investigational Site Number 2080003, Svendborg
- Investigational Site Number 2330001, Tallinn, Estonia
- France (6):
  - Investigational Site Number 2500005, Brest
  - Investigational Site Number 2500002, Montivilliers
  - Investigational Site Number 2500003, Montpellier
  - Investigational Site Number 2500007, Mulhouse
  - Investigational Site Number 2500001, Paris
  - Investigational Site Number 2500006, Pessac
- Germany (5):
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760002, Dresden
  - Investigational Site Number 2760003, Kirchheim unter Teck
  - Investigational Site Number 2760004, München
  - Investigational Site Number 2760007, Tübingen
- Investigational Site Number 3480001, Debrecen, Hungary
- Israel (2):
  - Investigational Site Number 3760006, Ashkelon
  - Investigational Site Number 3760004, Haifa
- Italy (2):
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800005, Rozzano
- Netherlands (4):
  - Investigational Site Number 5280005, Leeuwarden
  - Investigational Site Number 5280009, Sittard-Geleen
  - Investigational Site Number 5280007, The Hague
  - Investigational Site Number 5280001, Venlo
- Portugal (3):
  - Investigational Site Number 6200001, Almada
  - Investigational Site Number 6200005, Aveiro
  - Investigational Site Number 6200004, Ponte de Lima
- Russia (3):
  - Investigational Site Number 6430005, Kemerovo
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430003, Moscow
- Investigational Site Number 7050001, Ljubljana, Slovenia
- Spain (5):
  - Investigational Site Number 7240011, A Coruña
  - Investigational Site Number 7240010, Bilbao
  - Investigational Site Number 7240014, Madrid
  - Investigational Site Number 7240016, Sabadell
  - Investigational Site Number 7240015, Santa Cruz de Tenerife
- Sweden (2):
  - Investigational Site Number 7520003, Örebro
  - Investigational Site Number 7520001, Uppsala
- Investigational Site Number 7560002, Sankt Gallen, Switzerland
- United Kingdom (5):
  - Investigational Site Number 8260006, Aberdeen
  - Investigational Site Number 8260004, Gateshead
  - Investigational Site Number 8260003, Leeds
  - Investigational Site Number 8260005, Manchester
  - Investigational Site Number 8260011, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Schmidt WA, Dasgupta B, Sloane J, Giannelou A, Xu Y, Unizony SH, Mackie SL, Gonzalez-Gay MA, Spiera R, Warrington KJ, Villiger PM, Nivens MC, Akinlade B, Lin Y, Buttgereit F, Stone JH. A phase 3 randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of sarilumab in patients with giant cell arteritis. Arthritis Res Ther. 2023 Oct 16;25(1):199. doi: 10.1186/s13075-023-03177-6. PMID 37840134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 48 active centers in 19 countries. A total of 125 participants were screened between 20 November 2018 and 19 March 2020, of whom 42 participants were screen failures. Screen failures were mainly due to not meeting inclusion criteria. A total of 83 participants were enrolled and randomized in the study.
Pre-assignment Details: Participants were randomized to 4 treatments arms in 2:1:1:2 ratio by interactive response technology stratified by starting dose of prednisone at Baseline (less than [<] 30 milligrams per day (mg/day) or greater than or equal to [>=] 30 mg/day).
Groups:
- Sarilumab 150mg q2w+26 Week Taper: Participants received sarilumab 150 mg as SC injection q2w up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone-matching placebo from Week 26 up to Week 52.
- Sarilumab 200mg q2w+26 Week Taper: Participants received sarilumab 200 mg as SC injection q2w up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone-matching placebo from Week 26 up to Week 52.
Period: Overall Study
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Started | 28 | 14 | 14 | 27
Week 52 Analysis Set Population (Randomized participants who had opportunity to complete the 52-week treatment period (randomized prior to October 16th, 2019).) | 10 | 6 | 7 | 13
Completed | 9 | 6 | 6 | 8
Not Completed | 19 | 8 | 8 | 19
Not completed — Adverse Event | 2 | 1 | 1 | 7
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Other unspecified | 14 | 6 | 7 | 11

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper | Total Title
Number analyzed (Participants) | 28 | 14 | 14 | 27 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (7.7) | 69.5 (5.4) | 67.1 (7.9) | 73.4 (8.6) | 71.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 9 | 13 | 23 | 67
  Male | 6 | 5 | 1 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 23 | 13 | 11 | 25 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sustained Disease Remission at Week 52
Description: Disease remission was defined as resolution of signs and symptoms of giant cell arteries (GCA), and normalization of C-reactive protein (CRP) (<10 mg/L). Sustained remission was defined as meeting all of the following parameters: achievement of disease remission not later than Week 12, absence of disease flare (defined as recurrence of signs and symptoms attributable to active GCA plus an increase in corticosteroid [CS] dose due to GCA or elevation of erythrocyte sedimentation rate [ESR] attributable to active GCA plus an increase in CS dose due to GCA) from Week 12 through Week 52, normalization of CRP (to <10 mg/L, with absence of successive elevations to >=10 mg/L) from Week 12 through Week 52, and successful adherence to prednisone taper from Week 12 through Week 52.
Time Frame: At Week 52
Population: Analysis was performed on Week 52 analysis set population that included randomized participants who had opportunity to complete the 52-week treatment period (randomized prior to October 16th, 2019).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 7 | 13
percentage of participants | 30.0 | 0 | 42.9 | 46.2

2. Primary Outcome: Percentage of Participants Who Achieved Sustained Disease Remission at Week 24
Description: Disease remission was defined as resolution of signs and symptoms of GCA, and normalization of CRP <10 mg/L. Sustained remission was defined as meeting all of the following parameters: achievement of disease remission not later than Week 12, absence of disease flare (defined as recurrence of signs and symptoms attributable to active GCA plus an increase in CS dose due to GCA, or elevation of ESR attributable to active GCA plus an increase in CS dose due to GCA) from Week 12 through Week 24, normalization of CRP (to <10 mg/L, with an absence of successive elevations to >=10 mg/L) from Week 12 through Week 24, and successful adherence to the prednisone taper from Week 12 through Week 24.
Time Frame: At Week 24
Population: Analysis was performed on intent-to-treat (ITT) population that included participants who were allocated to a randomized treatment regardless of whether the treatment kit was used, and were analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
percentage of participants | 39.3 | 7.1 | 42.9 | 48.1

3. Secondary Outcome: Number of Participants With Achievement of Disease Remission up to Week 12: Week 52 Analysis Set
Description: Disease remission was defined as resolution of signs and symptoms of GCA, and normalization of CRP (< 10 mg/L). The status of normalization of CRP (<10 mg/L) was determined based on the last two non-missing post-baseline CRP values measured up to Week 12. If at least one of the value was <10 mg/L, then it was considered as normalization of CRP. Participants who took rescue corticosteroid (CS) due to active GCA prior to Week 12 or who permanently withdrew from the study treatment prior to Week 12 were considered as not achieved disease remission by Week 12.
Time Frame: Up to Week 12
Population: Analysis was performed on Week 52 analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 7 | 13
Participants | 7 | 3 | 4 | 7

4. Secondary Outcome: Number of Participants With Achievement of Disease Remission up to Week 12: Intent-to-treat (ITT) Population
Description: Disease remission was defined as resolution of signs and symptoms of GCA, and normalization of CRP (< 10 mg/L). The status of normalization of CRP (<10 mg/L) was determined based on the last two non-missing post-baseline CRP values measured up to Week 12. If at least one of the value was <10 mg/L, then it was considered as normalization of CRP. Participants who took rescue CS due to active GCA prior to Week 12 or who permanently withdrew from the study treatment prior to Week 12 were considered as not achieved disease remission by Week 12.
Time Frame: Up to Week 12
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
Participants | 16 | 6 | 9 | 15

5. Secondary Outcome: Number of Participants With Absence of Disease Flare From Week 12 Through Week 52: Week 52 Analysis Set
Description: Disease flare was defined as either recurrence of signs and symptoms attributable to active GCA plus an increase in CS dose due to GCA, or elevation of ESR attributable to active GCA plus an increase in CS dose due to GCA. Number of participants with absence of disease flare from Week 12 through Week 52 were reported.
Time Frame: From Week 12 through Week 52
Population: Analysis was performed on Week 52 analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 7 | 13
Participants | 7 | 3 | 4 | 7

6. Secondary Outcome: Number of Participants With Absence of Disease Flare From Week 12 Through Week 24: ITT Population
Description: Disease flare was defined as either recurrence of signs and symptoms attributable to active GCA plus an increase in CS dose due to GCA, or elevation of ESR attributable to active GCA plus an increase in CS dose due to GCA. Number of participants with absence of disease flare from Week 12 through Week 24 were reported.
Time Frame: From Week 12 through Week 24
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
Participants | 21 | 7 | 10 | 15

7. Secondary Outcome: Number of Participants With Normalization of C-Reactive Protein From Week 12 Through Week 52: Week 52 Analysis Set
Description: Normalization of CRP was defined as CRP levels <10 mg/L. If there were two or more consecutive visits with CRP >=10 mg/L, then it was categorized as no normalization of CRP.
Time Frame: From Week 12 through Week 52
Population: Analysis was performed on Week 52 analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 7 | 13
Participants | 6 | 3 | 5 | 8

8. Secondary Outcome: Number of Participants With Normalization of C-Reactive Protein (CRP) From Week 12 Through Week 24: ITT Population
Description: as for outcome 7
Time Frame: From Week 12 through Week 24
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
Participants | 20 | 4 | 11 | 17

9. Secondary Outcome: Number of Participants With Successful Adherence to the Prednisone Taper From Week 12 Through Week 52: Week 52 Analysis Set
Description: Successful adherence to the prednisone taper from Week 12 through Week 52 was defined as participants who did not take rescue therapy from Week 12 through Week 52 and might include the use of any excess prednisone (beyond the per protocol CS tapering regimen) with a cumulative dose of <=100 mg (or equivalent), such as those employed to manage adverse event (AE) not related to GCA.
Time Frame: From Week 12 through Week 52
Population: Analysis was performed on Week 52 analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 7 | 13
Participants | 6 | 2 | 3 | 6

10. Secondary Outcome: Number of Participants With Successful Adherence to the Prednisone Taper From Week 12 Through Week 24: ITT Population
Description: Successful adherence to the prednisone taper from Week 12 through Week 24 was defined as participants who did not take rescue therapy from Week 12 through Week 24 and might include the use of any excess prednisone (beyond the per protocol CS tapering regimen) with a cumulative dose of <=100 mg (or equivalent), such as those employed to manage AE not related to GCA.
Time Frame: From Week 12 through Week 24
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
Participants | 18 | 5 | 7 | 13

11. Secondary Outcome: Total Cumulative Corticosteroid (Including Prednisone) Dose
Description: Cumulative dose of CS used for GCA disease was defined as the dose taken up to the end of treatment, including expected prednisone in tapering regimen per protocol, CS used in rescue therapy and the use of commercial prednisone (an excess of <=100 mg of prednisone during the study treatment period employed to manage AE not related to GCA). The total cumulative CS dose was based on the total number of days with complete or partial intake, no imputation was done on missed tablets.
Time Frame: Up to Week 52
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
milligrams | 2577.3 (1018.3) | 2270.7 (1418.0) | 2177.1 (1326.7) | 1643.1 (967.3)

12. Secondary Outcome: Time to First Giant Cell Arteritis Disease Flare
Description: Time to first GCA flare was defined as the duration (in days) from randomization to first GCA flare after clinical remission (defined as resolution of signs and symptoms and normalization of CRP [<10 mg/L]) and up to 52 weeks. Disease flare was defined as either the recurrence of signs or symptoms attributable to active plus an increase in CS dose due to GCA or elevation of ESR attributable to active GCA plus an increase in CS dose due to GCA. Kaplan-Meier method was used for the analysis. Participants who never achieved remission were censored at randomization day; and those who achieved clinical remission and never flared were censored at the end of treatment assessment date up to Week 52.
Time Frame: Up to Week 52
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
days | NA [141.000 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to very low number of participants with the events. | 170.00 [85.000 to NA] — Upper limit of 95% CI was not estimable due to very low number of participants with the events. | NA [58.000 to NA] — Median and upper limit of 95% CI was not estimable due to very low number of participants with the events. | NA [77.000 to NA] — Median and upper limit of 95% CI was not estimable due to very low number of participants with the events.

13. Secondary Outcome: Composite Glucocorticoid Toxicity Index (C-GTI): Cumulative Worsening Score (CWS) and Aggregate Improvement Score (AIS) at Week 24: ITT Population
Description: GTI assessed glucocorticoid (GC) related morbidity and GC-sparing ability of other therapies; composed of 2 components: Composite GTI and Specific List. Composite GTI contained 9 domains and Specific List contained of 23 items (11 domains), used as complementary tool to C-GTI. Composite GTI score was the sum of 9 domain-specific scores at each visit and Cumulative GTI score was the sum of composite GTI scores across each visit. Two cumulative GTI scores: CWS and AIS at Week 24 are reported in this outcome measure (OM). CWS assessed cumulative GC toxicity regardless of whether toxicity had lasting effects or was transient. AIS assessed new therapy effectiveness in decreasing any Baseline GC toxicity over time. For CWS, composite score ranged from 0 to 439 and for AIS, composite score ranged from -346 to 439. For both CWS and AIS, the minimum score implies the least toxicity and the maximum score implies the most toxicity.
Time Frame: At Week 24
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
units on a scale
  Cumulative worsening score | 29.2 (30.8) | 30.7 (33.2) | 55.1 (43.1) | 31.0 (42.9)
  Aggregate improvement score | -21.6 (54.8) | -13.4 (44.3) | 14.2 (55.0) | -3.3 (43.4)

14. Secondary Outcome: Composite Glucocorticoid Toxicity Index: Cumulative Worsening Score and Aggregate Improvement Score at Week 52
Description: GTI assessed glucocorticoid (GC) related morbidity and GC-sparing ability of other therapies; composed of 2 components: Composite GTI and Specific List. Composite GTI contained 9 domains and Specific List contained of 23 items (11 domains), used as complementary tool to C-GTI. Composite GTI score was the sum of 9 domain-specific scores at each visit and Cumulative GTI score was the sum of composite GTI scores across each visit. Two cumulative GTI scores: CWS and AIS at Week 52 are reported in this OM. CWS assessed cumulative GC toxicity regardless of whether toxicity had lasting effects or was transient. AIS assessed new therapy effectiveness in decreasing any Baseline GC toxicity over time. For CWS, composite score ranged from 0 to 439 and for AIS, composite score ranged from -346 to 439. For both CWS and AIS, the minimum score implies the least toxicity and the maximum score implies the most toxicity.
Time Frame: At Week 52
Population: Analysis was performed on Week 52 analysis set. Here, 'overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 10 | 6 | 6 | 11
units on a scale
  Cumulative worsening score | 73.0 (50.3) | 84.7 (33.4) | 77.2 (41.7) | 52.8 (39.0)
  Aggregate improvement score | -19.5 (65.0) | 31.2 (54.7) | 23.7 (31.9) | -0.5 (51.5)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious AEs (SAEs) were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were the AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the investigational medicinal product (IMP) to the last dose of the SC IMP +60 days).
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose (i.e., up to Week 60)
Population: Analysis was performed on safety population that included participants who had received at least one dose or part of a dose of IMP and were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
Participants
  Any TEAE | 24 | 14 | 13 | 22
  Any treatment emergent SAE | 2 | 3 | 2 | 7

16. Secondary Outcome: Pharmacokinetics (PK): Serum Trough Concentration (Ctrough) of Sarilumab
Description: Ctrough was pre dose concentration of drug. Data for this outcome measure was not planned to be collected and analyzed for placebo arms (Placebo+52 Week Taper and Placebo+26 Week Taper) as pre-specified in the protocol.
Time Frame: Pre-dose on Week 0 (Baseline), Weeks 2, 4, 12, 16, 24 and 52
Population: Analyzed on PK analysis population: participants who had received at least one dose or part of a dose of IMP, were analyzed according to the treatment actually received and had at least 1 post-dose non-missing serum sarilumab concentration value. Here, 'Number Analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 14 | 26
nanograms per milliliter
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 14 | 25
  Week 2 | 2099.29 (3114.92) | 5400.82 (4124.63)
  Week 4: number analyzed (Participants) | 13 | 25
  Week 4 | 4644.71 (5994.17) | 11640.98 (8574.00)
  Week 12: number analyzed (Participants) | 13 | 20
  Week 12 | 8371.33 (7608.42) | 27586.00 (17496.07)
  Week 16: number analyzed (Participants) | 12 | 17
  Week 16 | 8111.08 (5962.56) | 28911.88 (20821.06)
  Week 24: number analyzed (Participants) | 12 | 19
  Week 24 | 12926.67 (9509.92) | 35451.74 (23953.29)
  Week 52: number analyzed (Participants) | 6 | 9
  Week 52 | 19780.00 (21829.95) | 46766.67 (21172.15)

17. Secondary Outcome: Pharmacokinetics: Serum Drug Concentration of Sarilumab Post-dose at Week 24
Description: Serum concentrations of functional sarilumab were analyzed using validated enzyme linked immunosorbent assay.
Time Frame: post-dose at Week 24
Population: Analysis was performed on PK analysis population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for placebo arms (Placebo+52 Week Taper and Placebo+26 Week Taper) as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 11 | 13
nanograms per milliliter | 25255.45 (17510.38) | 44551.54 (28298.62)

18. Secondary Outcome: Percentage of Participants With Treatment-emergent Antidrug Antibodies (ADA) Response
Description: ADA response categories: 1) Treatment-boosted ADA positive participant: Participant with a positive ADA assay response at Baseline and with at least a 4-fold increase in titer compared to Baseline during TEAE period. 2) Treatment-emergent ADA positive participant: Participant with non-positive assay (meaning negative or missing) response at Baseline but with a positive assay response during the TEAE period (defined as the time from the first dose of the IMP to the last dose of the SC IMP + 60 days). Titer values were categorized as low (titer <1,000); moderate (1,000<= titer <=10,000) and high (titer >10,000).
Time Frame: From Day 1 (Baseline) up to last dose date of study drug + 60 days (i.e., up to Week 60)
Population: Analysis was performed on ADA population that included participants who had received at least one dose or part of a dose of IMP, were analyzed according to the treatment actually received and had at least 1 non-missing ADA result in the ADA assay following the first dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 26 | 13 | 14 | 24
percentage of participants
  Treatment-boosted ADA positive participants | 0 | 0 | 0 | 0
  Treatment-emergent ADA positive participants | 3.8 | 0 | 7.1 | 0

19. Secondary Outcome: Pharmacodynamics: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 52
Description: ESR is a laboratory test to provide non-specific measure of inflammation in the body. The test assessed the rate at which red blood cells fell in a test tube and was measured in millimeters per hour.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: Analysis was performed on ITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: millimeters per hour
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
millimeters per hour
  Baseline: number analyzed (Participants) | 28 | 13 | 14 | 27
  Baseline | 29.3 (27.3) | 21.9 (16.2) | 24.9 (22.0) | 18.2 (16.8)
  Week 2: number analyzed (Participants) | 27 | 11 | 14 | 24
  Week 2 | -1.1 (17.9) | 0.7 (11.4) | -10.4 (16.4) | -8.8 (12.4)
  Week 4: number analyzed (Participants) | 25 | 10 | 13 | 25
  Week 4 | -4.2 (21.4) | 5.2 (19.7) | -13.3 (22.6) | -9.4 (15.2)
  Week 8: number analyzed (Participants) | 24 | 13 | 12 | 24
  Week 8 | -2.0 (22.7) | 10.2 (12.6) | -11.9 (18.9) | -8.7 (16.1)
  Week 12: number analyzed (Participants) | 21 | 13 | 12 | 23
  Week 12 | -1.5 (24.9) | 9.8 (13.3) | -14.7 (19.2) | -11.0 (14.1)
  Week 16: number analyzed (Participants) | 22 | 12 | 13 | 19
  Week 16 | -4.1 (22.7) | 9.8 (16.5) | -13.5 (18.1) | -10.4 (12.7)
  Week 20: number analyzed (Participants) | 21 | 11 | 14 | 20
  Week 20 | -6.6 (23.7) | 8.8 (14.6) | -18.2 (23.5) | -10.9 (12.2)
  Week 24: number analyzed (Participants) | 21 | 10 | 14 | 22
  Week 24 | -4.2 (22.0) | 13.9 (16.1) | -16.4 (25.6) | -9.3 (11.5)
  Week 32: number analyzed (Participants) | 22 | 10 | 9 | 17
  Week 32 | -7.0 (21.3) | 6.6 (16.2) | -9.4 (18.0) | -7.9 (10.6)
  Week 40: number analyzed (Participants) | 19 | 8 | 8 | 14
  Week 40 | -1.5 (22.3) | 4.0 (18.1) | -10.1 (25.2) | -7.9 (8.6)
  Week 52: number analyzed (Participants) | 13 | 7 | 6 | 10
  Week 52 | -1.0 (27.0) | -1.4 (12.4) | -15.2 (19.0) | -7.0 (12.0)

20. Secondary Outcome: Pharmacodynamics: Change From Baseline in C-reactive Protein (CRP) Level at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 52
Description: CRP is a protein made by the liver. CRP levels increase in blood when inflammation occurs in the body.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 52
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
milligrams per liter
  Baseline | 10.9 (20.0) | 9.7 (18.3) | 10.1 (12.4) | 3.7 (6.2)
  Week 2: number analyzed (Participants) | 26 | 11 | 14 | 26
  Week 2 | 0.4 (21.0) | -1.0 (21.2) | -3.5 (11.2) | -2.0 (7.6)
  Week 4: number analyzed (Participants) | 25 | 11 | 13 | 25
  Week 4 | -3.6 (19.3) | -2.2 (21.8) | -2.6 (18.7) | -1.9 (8.3)
  Week 8: number analyzed (Participants) | 23 | 12 | 12 | 21
  Week 8 | -4.0 (19.5) | -0.9 (17.0) | -3.5 (11.7) | -1.7 (5.5)
  Week 12: number analyzed (Participants) | 21 | 12 | 13 | 21
  Week 12 | -4.4 (22.0) | 4.4 (18.9) | -3.3 (17.9) | -1.1 (8.4)
  Week 16: number analyzed (Participants) | 22 | 11 | 13 | 16
  Week 16 | -4.5 (20.7) | 5.0 (23.9) | -5.0 (14.1) | -1.8 (3.0)
  Week 20: number analyzed (Participants) | 21 | 9 | 13 | 18
  Week 20 | -4.5 (21.1) | 0.6 (17.6) | -4.9 (13.6) | -1.6 (2.9)
  Week 24: number analyzed (Participants) | 21 | 7 | 12 | 18
  Week 24 | -4.1 (19.5) | 0.3 (32.6) | -3.1 (18.3) | -1.0 (4.5)
  Week 32: number analyzed (Participants) | 21 | 7 | 7 | 14
  Week 32 | -5.2 (19.6) | 1.1 (35.4) | -5.8 (17.1) | -0.4 (6.5)
  Week 40: number analyzed (Participants) | 16 | 6 | 7 | 10
  Week 40 | -1.9 (22.3) | -9.2 (27.0) | -2.2 (11.1) | -2.8 (3.5)
  Week 52: number analyzed (Participants) | 7 | 4 | 4 | 5
  Week 52 | 8.2 (27.4) | -13.8 (37.0) | -4.5 (5.2) | -4.6 (4.4)

21. Secondary Outcome: Pharmacodynamics: Change From Baseline in Interleukin-6 (IL-6) at Weeks 2, 12, 24, and 52
Description: Interleukin-6 is a protein produced in the body. Levels of IL-6 often increase when there is inflammation (redness, warmth, swelling, and pain as a result of infection, irritation, or injury), either acute or chronic.
Time Frame: Baseline, Weeks 2, 12, 24, and 52
Population: Analysis was performed on safety population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per Liter
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
nanograms per Liter
  Baseline: number analyzed (Participants) | 25 | 12 | 13 | 23
  Baseline | 10.91 (12.85) | 8.74 (5.78) | 11.03 (15.33) | 7.71 (7.30)
  Week 2: number analyzed (Participants) | 23 | 8 | 13 | 22
  Week 2 | 2.90 (17.46) | 3.47 (10.30) | 31.74 (31.13) | 117.33 (245.28)
  Week 12: number analyzed (Participants) | 18 | 7 | 11 | 17
  Week 12 | -0.88 (12.60) | 5.56 (8.08) | 52.38 (47.46) | 81.82 (50.85)
  Week 24: number analyzed (Participants) | 20 | 4 | 11 | 15
  Week 24 | -1.03 (7.15) | 5.57 (19.81) | 53.60 (53.71) | 69.20 (46.89)
  Week 52: number analyzed (Participants) | 7 | 3 | 3 | 6
  Week 52 | 0.43 (5.58) | 2.82 (1.90) | 42.14 (8.52) | 33.28 (32.37)

22. Secondary Outcome: Pharmacodynamics: Change From Baseline in Soluble Interleukin-6 Receptor (sIL-6R) Level at Weeks 2, 12, 24, and 52
Description: Interleukin-6 is a protein produced in the body. Levels of IL-6 often increase when there is inflammation (redness, warmth, swelling, and pain as a result of infection, irritation, or injury), either acute or chronic. sIL-6R is one of the receptors that bind IL-6.
Time Frame: Baseline, Weeks 2, 12, 24, and 52
Population: Analyzed on safety population. Here, 'Number Analyzed'=participants with available data for each specified category and '0' in number analyzed field signifies that no participants were available for assessments at specified time points in the respective arm.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
Number analyzed (Participants) | 28 | 14 | 14 | 27
nanograms per milliliter
  Baseline: number analyzed (Participants) | 27 | 14 | 13 | 27
  Baseline | 136.63 (260.57) | 54.80 (18.48) | 50.05 (17.84) | 61.37 (72.43)
  Week 2: number analyzed (Participants) | 0 | 0 | 13 | 26
  Week 2 |  |  | 212.19 (51.99) | 224.87 (107.43)
  Week 12: number analyzed (Participants) | 1 | 0 | 12 | 21
  Week 12 | 17.67 |  | 336.30 (107.49) | 427.40 (124.97)
  Week 24: number analyzed (Participants) | 3 | 0 | 11 | 18
  Week 24 | -12.72 (3.97) |  | 311.88 (184.32) | 456.09 (118.07)
  Week 52: number analyzed (Participants) | 8 | 2 | 4 | 7
  Week 52 | -131.47 (356.65) | -9.69 (11.14) | 377.23 (84.99) | 471.16 (182.72)

ADVERSE EVENTS:
Time Frame: From first dose (i.e., Day 1) of study drug to last dose date of study drug + 60 days (i.e., up to Week 60)
Description: Reported AEs and deaths were treatment emergent AEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of the IMP to the last dose of the SC IMP + 60 days). Analysis was performed on safety population.
Arm/Group | Placebo+52 Week Taper | Placebo+26 Week Taper | Sarilumab 150mg q2w+26 Week Taper | Sarilumab 200mg q2w+26 Week Taper
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/14 | 0/14 | 2/27
Serious Adverse Events (participants affected / at risk) | 2/28 | 3/14 | 2/14 | 7/27
Other Adverse Events (participants affected / at risk) | 22/28 | 13/14 | 13/14 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+52 Week Taper (N=28) | Placebo+26 Week Taper (N=14) | Sarilumab 150mg q2w+26 Week Taper (N=14) | Sarilumab 200mg q2w+26 Week Taper (N=27)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blindness Unilateral (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Amyloid Angiopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic Dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+52 Week Taper (N=28) | Placebo+26 Week Taper (N=14) | Sarilumab 150mg q2w+26 Week Taper (N=14) | Sarilumab 200mg q2w+26 Week Taper (N=27)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amaurosis Fugax (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Cataract Subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Refraction Disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 2 (2) | 3 (3) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection Site Rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 4 (8) | 1 (1)
Injection Site Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vessel Puncture Site Phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaccination Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine Renal Clearance Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Steroid Diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning Sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Decreased Vibratory Sense (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (7) | 1 (1) | 4 (5)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Mania (Psychiatric disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (2)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Fragility (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was prematurely discontinued due to protracted enrolment exacerbated by Covid-19 pandemic situation and not due to any safety issues from administration of sarilumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03600805/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03600805/SAP_001.pdf